CLINICAL TRIAL: NCT04929457
Title: Evaluation of Digiphysical Screening for Familial Hypercholesterolemia - Efficacy of Digiphysical Screening, Effects on Cardiovascular Morbidity and Mortality and Health Economic Aspects
Brief Title: Evaluation of a Digiphysical Screening Method to Identify and Diagnose Familial Hypercholesterolemia
Acronym: DigiLipids
Status: Enrolling by invitation | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jonas Brinck, Principal Investigator, Karolinska Institutet
Other Study IDs: DigiLipids
Record Dates: First submitted 2021-05-28; First posted 2021-06-18 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Familial Hypercholesterolemia; Hypercholesterolemia
Keywords: familial hypercholesterolemia; cardiovascular disease; coronary artery disease; ischemic stroke; peripheral artery disease; hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia; Cardiovascular Diseases; Coronary Artery Disease; Ischemic Stroke; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals screened for Familial Hypercholesterolemia: Individuals participating in diagnostic activities in the digiphysical health care screening program for Familial Hypercholesterolemia and have provided informed consent are included in the cohort.

SUMMARY:
Longitudinal and observational registry-based cohort study of individuals participating in the national digiphysical screening program for Familial Hypercholesterolemia. The information collected in the screening process will be combined in pseudo-anonymous form with data from the National Board of Health and Welfare (registries: Cause of Death, Diagnoses according to International Classification of Diseases (ICD) and Prescribed drugs) and Statistic Sweden (Longitudinal integrated database for health insurance and labour market studies). Primary analysis: association between Familial Hypercholesterolemia and cardiovascular disease. Secondary analysis: efficacy and health economic aspects of digiphysical screening for Familial Hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Swedish personal identification number

Exclusion Criteria:

* Decline informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals that partake in the Swedish national digiphysical screening program for Familial Hypercholesterolemia will be asked to give personal informed consent to participate in the longitudinal observational cohort study.
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease burden in patients with newly diagnosed Familial Hypercholesterolemia | Through study completion, until 2041.
  Presence of ischemic heart disease, ischemic cerebrovascular disease and/or peripheral artery disease in relation to age in patients with newly diagnosed Familial Hypercholesterolemia. Data is reported after 2, 5, 10, 15 and 20 years.
Change in cardiovascular disease burden in patients with diagnosed Familial Hypercholesterolemia | Through study completion, until 2041.
  Change in presence of ischemic heart disease, ischemic cerebrovascular disease and/or peripheral artery disease in relation to age in patients diagnosed Familial Hypercholesterolemia. Comparison is done between baseline and after 2, 5, 10, 15 and 20 years.
Impact of mutation positive Familial Hypercholesterolemia on cardiovascular disease burden | Through study completion, until 2041.
  Comparison of cardiovascular disease burden (presence of ischemic heart disease, ischemic cerebrovascular disease and/or peripheral artery disease) in relation to age in patients with mutation positive versus negative Familial Hypercholesterolemia. Data is reported after 2, 5, 10, 15 and 20 years.
Comparison of cardiovascular disease burden between patients with diagnosed Familial Hypercholesterolemia and individuals aquitted from the diagnose | Through study completion, until 2041.
  Comparison of cardiovascular disease burden (presence of ischemic heart disease, ischemic cerebrovascular disease and/or peripheral artery disease) in relation to age between patients diagnosed with Familial Hypercholesterolemia and individuals screened but acquitted of the diagnose.
  Data is reported after 2, 5, 10, 15 and 20 years.

SECONDARY OUTCOMES:
Key efficacy numbers and ratios of screened and diagnosed for the digiphysical screening method to diagnose Familial Hypercholesterolemia | Through study completion, until 2041.
  The efficacy of the digiphysical screening method will be assessed by key numbers and ratios:
  * screened
  * biochemically tested with cholesterol measurement
  * genetically tested
  * diagnosed with Familial Hypercholesterolemia
  * biochemically tested/screened
  * genetically tested/screened
  * diagnosed with Familial Hypercholesterolemia/screened
  Data is reported after 2, 5, 10, 15 and 20 years.
Health economic aspects of the digiphysical screening method to diagnose Familial Hypercholesterolemia | Through study completion, until 2041.
  Costs and cost-benefits for digiphysical screening and treatment of individuals diagnosed with Familial Hypercholesterolemia.
  Data is reported after 2, 5, 10, 15 and 20 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Brinck, MD PhD, Principal Investigator — Dept. of Medicine Huddinge H7, Karolinska Institute, Stockholm
Locations (1):
- Karolinska university hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request data sharing is possible after discussion with responsible researchers.
Time Frame: First result anticipated two years after start.
Access Criteria: Ethical committee approval Purpose to publish results in peer-reviewed international scientific journal